CLINICAL TRIAL: NCT03911765
Title: Effect of Digital Cognitive Training on the Functionality of Older Adults With Mild Cognitive Impairment (MCI)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rogerio Panizzutti, Director, Clinical Research, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17976113.1.0000.5257
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Stepped wedge
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Executive Function cognitive training (Experimental): 20 hours of digital cognitive training targeting executive function.
  Interventions: Behavioral: digital cognitive training
- Games (Active Comparator): 10 hours of computer games c available online which do not involve a high demand in cognitive functions (e.g. fishing game, pinball game, tetris, etc), followed by 10 hours of of digital cognitive training targeting executive function.
  Interventions: Behavioral: digital cognitive training

INTERVENTIONS:
Behavioral: digital cognitive training — Digital cognitive exercises, used in the intervention group, have the primary objective of stimulating executive functions, and will be made available through the Internet using the BrainHQ platform.

SUMMARY:
The purpose of this study is to investigate the effect of digital cognitive training in the functionality of older adults with Mild Cognitive Impairment.

DETAILED DESCRIPTION:
Mild Cognitive Impairment (MCI) is characterized by decline in one or more cognitive domains, including memory, attention, executive functions, language and visuospatial abilities, and in a significant portion of cases may evolve to Alzheimer's Disease. According to established diagnostic criteria, independence for daily life activities is preserved, but activities are carried out less effectiveness and efficiency, affected subjects usually take more time and make more mistakes, when compared to their pre-morbid performance. Different studies have observed that impairments in functional performance in older adults with MCI are associated with impairments in executive function. This study intends to verify the impact of the use of digital cognitive training for executive function on the functionality of older adults with MCI. Digital cognitive exercises, used in the intervention group, have the primary objective of stimulating executive functions, and will be made available through the Internet using the BrainHQ platform. The active control group will play computer games available online. Both groups will play for 1 hour at least 2 times per week.

After baseline assessments, older adults with MCI will be stratified by age, education, gender, functional measurement and cognitive assessment, and randomly assigned to the intervention group with digital cognitive exercises or to the control group with computer games, in a stepped wedge design. Subjects will be evaluated at baseline and after completing 10 and 20 hours of intervention. After the first 10 hours of intervention both groups will be assigned to the intervention with digital cognitive exercises for additional 10 hours. Both groups will be comparable in terms of personal contact with staff and computer time. Our hypothesis is that the training using digital cognitive exercises will improve the executive function and that this gain has a positive impact on the functionality and accomplishment of the daily life activities of older adults with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 years old;
* Elderly enrolled in home for aged in wich the research is taking place;
* Montreal Cognitive Assessment above 21 points;

Exclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease;
* Serious medical or neurological condition preventing from participation in the study;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-02 (Estimated)

PRIMARY OUTCOMES:
Performance in everyday living score change | 3 months
  Performance in everyday living score change will be measured using Canadian Occupational Performance Measure (COPM).
  The Canadian Occupational Performance Measure (COPM) has a client-centered design and measures outcomes according to three occupational performance areas (self-care, productivity, and leisure), examining self-perceived changes in the occupational performance of patients through a semistructured interview. At the beginning, patients start by identifying their difficulties according to the three occupational performance areas. They subsequently use a 10-point scale, ranging from not at all crucial (1) to extremely crucial (10), to identify the intensity of certain difficulties. For the top five problems or tasks selected by patients, the interviewer asks them to continue identifying their performance and satisfaction with their performance by using the same 10-point rating scale.

SECONDARY OUTCOMES:
Functional status score change | 3 months
  Functional status score will be measured using the Direct Assessment of Functional Status-Revised (DAFS-R). DAFS-R assesses seven different domains of functional abilities by requiring the participant to carry out different tasks, two domains will be evaluated: dealing with Finances (score range 0-32) and shopping skills (score range 0-20), with higher scores indicating better functioning.

OTHER OUTCOMES:
Global cognitive function score change | 3 months
  Global cognitive function score will be measured using the Montreal Cognitive Assessment (MoCA). Thirty items assessing multiple cognitive domains are contained in the MoCA: short-term memory (score range 0-5); visuospatial abilities (score range 0-3), cube copy task (score range 0-1); executive functioning (score range 0-1), phonemic fluency (score range 0-1), verbal abstraction (score range 0-2); attention, concentration, and working memory (score range 0-1), serial subtraction (score range 0-3), digits forward (score range 0-1), and digits backward (score range 0-1); language (score range 0-3), and repetition of complex sentences (score range 0-2); orientation to time and place (score range 0-6), with higher scores indicating better cognition.
Semantic memory score change | 3 months
  Semantic memory score will be measured using the Verbal fluency test. The verbal fluency test is a short test of verbal functioning. It typically consists of two tasks: category fluency and letter fluency. In the standard versions of the tasks, participants are given 1 min to produce as many unique words as possible within a semantic category (category fluency) or starting with a given letter (letter fluency). The participant's score in each task is the number of unique correct words.
Selective attention and cognitive flexibility | 3 months
  Selective attention and cognitive flexibility will be measured using the Stroop Test
Sustained attention and set-shifting | 3 months
  Sustained attention and set-shifting will be measured using the Trial Making Test
Depression score change | 3 months
  Depression score will be measured using the Geriatric Depression Scale - 15 (Short version). The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly. In the Geriatric Depression Scale, questions are answered "yes" or "no." One point is assigned to each answer and the cumulative score is rated on a scoring grid. The grid sets a range of 0-9 as "normal", 10-19 as "mildly depressed", and 20-30 as "severely depressed".
Qualitative motivation with the computerized training exercise | 3 months
  Qualitative motivation will be assessed using semi-structured interview

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro, Brazil